CLINICAL TRIAL: NCT00104468
Title: An Open-Label, Single-Arm, Multi-Center, Phase I Study of Troxatyl™ (Troxacitabine) Administered by Continuous Infusion in Subjects With Refractory Acute Myelogenous Leukemia
Brief Title: Study of Troxatyl™ Administered by Continuous Infusion to Subjects With Refractory Acute Myelogenous Leukemia (AML)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Trial stopped June 2007
Sponsor: SGX Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD758-110
Record Dates: First submitted 2005-02-28; First posted 2005-03-01 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Single-arm, open-label, multi-center, dose escalation, continuous infusion, multi-dose, acute myeloid leukemia; Acute myelogenous leukemia (AML) that has been refractory to prior therapy and/or is unlikely to benefit from known therapies
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — troxacitabine

INTERVENTIONS:
Drug: Troxatyl™ (Cytotoxic Chemotherapeutic)

SUMMARY:
This is a phase I, single-arm, open-label, multi-center study of rising doses of Troxatyl™ whose purpose is to determine the safety, tolerance, and pharmacokinetics, and to establish the recommended infusion schedule of Troxatyl™.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of acute myelogenous leukemia (AML) refractory to prior therapy and/or unlikely to benefit from known therapies.
* Subjects must have adequate organ and immune function as indicated by the following laboratory values: *Creatinine clearance ≥5 L/hr (83mL/min), *Total Bilirubin ≤2.0 mg/dL (≤34.2 µmol/L), *AST(SGOT) and ALT(SGPT) ≤3 x ULN

Exclusion Criteria:

* Clinical evidence of active central nervous system (CNS) leukemic involvement
* Active and uncontrolled infection
* Uncontrolled medical problems unrelated to the malignancy that impair their ability to give informed consent or unacceptably reduce the safety of the proposed treatment
* Neurologic or psychiatric disorders that would interfere with informed consent or study follow-up
* Known or suspected intolerance or hypersensitivity to the investigational new drug or closely related compounds like lamivudine, and/or a recent history of alcohol or other substance abuse.
* Also not eligible are subjects who have used another investigational agent or participated in a clinical trial within the last 14 days prior to enrollment.
* Females with a positive pregnancy test at screening or subjects that have previously been enrolled into this study and subsequently withdrew.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To determine the recommended infusion schedule for the investigational new drug administered as a continuous infusion with regards to dose limiting toxicities.

SECONDARY OUTCOMES:
Pharmacokinetic/pharmacodynamic profile, preliminary evidence of the anti-tumor activity.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cornell Medical College, New York Presbyterian, New York, New York
  - MD Anderson, Houston, Texas

REFERENCES:
- [Background] Giles FJ. Troxacitabine-based therapy of refractory leukemia. Expert Rev Anticancer Ther. 2002 Jun;2(3):261-6. doi: 10.1586/14737140.2.3.261. PMID 12113049